CLINICAL TRIAL: NCT04984408
Title: A Phase 3, Randomized, Observer-blind, Controlled Trial to Assess the Efficacy, Immunogenicity and Safety of BBIBP-CorV Vaccine Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Brief Title: Efficacy, Immunogenicity and Safety of BBIBP-CorV Vaccine Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection.
Acronym: ECOVA-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IVI-ECOVA-01
Record Dates: First submitted 2021-07-28; First posted 2021-07-30 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Disease

STUDY DESIGN:
Intervention Model Description: A randomized, observer-blind, controlled, phase 3 trial will be conducted to assess the safety, immunogenicity and efficacy of two doses of intramuscular BBIBP-CorV vaccine, followed by a booster dose, in adults 18 years of age and older.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The PI, study staff, and participants will be blinded as to receipt of study vaccine or comparator. The pharmacy staff preparing the vaccine syringes and the study nurse who is administering the vaccine will not be involved in the safety assessment of participants and will be instructed not to comment on the experimental agent to study staff. Enrollment numbers will be assigned sequentially by the study nurse/pharmacist upon confirmation of eligibility and enrollment into the study according to their Human Immunodeficiency Virus (HIV) stratification by the Investigator. All case report forms (CRFs) and source documents will be labeled with the enrollment number and study visit number. Personal identifying information linking the study number to an individual volunteer will not be captured on case report form (CRF) as study data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: BBIBP-CorV (Experimental): Study Arms 1 will have two groups: group 1 - HIV-uninfected receiving BBIBP-CorV; group 2 - HIV-infected receiving BBIBP-CorV .
  Interventions: Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell)
- Arm 2: Flu Quadrivalent (Experimental): Study Arms 2 will have two groups: group 1 - HIV-uninfected receiving Flu Quadrivalent; group 2 - HIV-infected receiving Flu Quadrivalent. The Flu Quadrivalent is recommended as a single dose for adults, the second and the booster doses for Arm 2 will be placebo.
  Interventions: Biological: influenza season quadrivalent Influenza Vaccine (Flu Quadrivalent)
- Arm 3: BBIBP-CorV and Flu Quadrivalent (Co-administration) (Experimental): Arm 3 will have 1 group - HIV-uninfected co-administration group receiving both study vaccines.
  Interventions: Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell); Biological: influenza season quadrivalent Influenza Vaccine (Flu Quadrivalent)

INTERVENTIONS:
Biological: BBIBP-CorV - Inactivated SARS-CoV-2 vaccine (Vero cell) — * The Inactivated SARS-CoV-2 vaccine (Vero cell)- BBIBP-CorV manufactured by Beijing Institute of Biological Products (BIBP), China National Biotec Group (CNBG), Sinopharm, Beijing, People's Republic of China
  * Dose formulation: A liquid formulation containing 4μg total protein with aluminum hydroxide adjuvant (0·45 mg/mL) per 0·5 mL (2-dose schedule followed by a booster dose).
  * Mode of Administration: Intramuscular
  * Storage Conditions: 2 to 8 degree Celsius
  Arms: Arm 1: BBIBP-CorV; Arm 3: BBIBP-CorV and Flu Quadrivalent (Co-administration)
Biological: influenza season quadrivalent Influenza Vaccine (Flu Quadrivalent) — * The southern hemisphere for the 2021 influenza season quadrivalent Influenza Vaccine (Flu Quadrivalent)
  * Dose formulation: Purified Inactivated Influenza Virus Antigen H1N1, H3N2, Yamagata and Victoria (single dose, 0.5ml for adults)
  * Mode of Administration: Intramuscular
  * Storage Conditions: 2 to 8 degree Celsius
  Arms: Arm 2: Flu Quadrivalent; Arm 3: BBIBP-CorV and Flu Quadrivalent (Co-administration)

SUMMARY:
To expand the access and delivery of COVID-19 Vaccines in Africa (ECOVA), the investigators will conduct a phase 3, individually randomized, observer-blind, controlled (influenza vaccine) trial to evaluate the safety and efficacy of the BBIBP-CorV vaccine against any severe acute respiratory syndrome 2 (SARS-CoV- 2) infection among adults 18 years and older. The BBIBP-CorV vaccine is an inactivated SARS-CoV-2 vaccine (Vero cell) manufactured by the Beijing Institute of Biological Products (BIBP), China National Biotec Group (CNBG), Sinopharm, Beijing, People's Republic of China and received emergency use authorization (EUA) from World Health Organization (WHO).

DETAILED DESCRIPTION:
The investigators will conduct a randomized, observer-blind, controlled, phase 3 trial will be conducted to assess the safety, immunogenicity and efficacy of two doses of intramuscular BBIBP-CorV vaccine, followed by a booster dose, in adults 18 years of age and older. . Study Arms 1 and 2 will have two groups: group 1 - HIV-uninfected receiving BBIBP-CorV or Flu Quadrivalent; group 2 - HIV-infected receiving BBIBP-CorV or Flu Quadrivalent. Arm 3 will have 1 group - HIV-uninfected co-administration group receiving both vaccines. The randomization will be stratified by HIV status. Active surveillance for covid-19 will be carried out and immunogenicity will be assessed for a subset of population.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adults aged 18 years and older (Arm 1-Group 1 and Arm 2-Group 1) and 18-65 years (Arm 1 - Group 2, Arm 2-Group 2 and Arm3-Group1) at the time of consent.
* Residing within the Beira and Maputo health region and planning to stay for the study duration.
* HIV-negative test result at the day of screening for participants in Group 1, in Arms 1, 2 and 3
* HIV-positive and on anti-retroviral treatment for at least six months for participants in Group 2, in Arms 1 and 2
* Female volunteers of childbearing potential with a negative pregnancy test on the day(s) of screening and vaccination, practicing/willing to practice continuous effective contraception recommended by the national health system up to four weeks after the third vaccination.
* Able and willing to comply with all study requirements, based on the assessment of the investigator.
* Provide written informed consent before any trial procedure.

Exclusion Criteria:

* Pregnant, lactating, or with intention to become pregnant during the study.
* Planned receipt of any investigational vaccine than the study intervention within 28 days before and after each study vaccination.
* Active COVID-19 infection at the time of enrollment
* History of allergic reactions or anaphylaxis to previous immunization or allergies to any components of the vaccines.
* History of bleeding disorder, or prior history of significant bleeding or bruising following intramuscular injections or venipuncture (for the immunogenicity subset and HIV infected participants).
* Any other finding which in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial or result in incomplete or poor quality data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8825 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Protection conferred by BBIBP-CorV vaccine against any COVID-19 disease | Up to two years follow up from the date of enrollment
  Protection conferred by BBIBP-CorV vaccine against any COVID-19 disease measured as the reduction in incidence of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) confirmed COVID-19 disease in the BBIBP-CorV vaccine arm (s) compared to the control arm, 7 days after the second dose of study intervention

SECONDARY OUTCOMES:
Incidence of solicited adverse events, unsolicited adverse events and serious adverse events and adverse events of special interest (AESIs) | local solicited adverse events within 7 days and systemic solicited adverse events within 14 days of each vaccination, unsolicited adverse events within 28 days of each vaccination
  Incidence of local solicited adverse events within 7 days and systemic solicited adverse events within 14 days of each vaccination, unsolicited adverse events within 28 days of each vaccination, serious adverse events and adverse events of special interest (AESIs) throughout the duration of the study according to the Brighton collaboration list for COVID-19 vaccine studies
Protection conferred by BBIBP-CorV vaccine against symptomatic COVID-19 disease | Till two years follow up from the date of enrollment
  Protection conferred by BBIBP-CorV vaccine against symptomatic COVID-19 disease caused by variants of concerns (VoCs) measured as the reduction in incidence of RT-PCR-confirmed symptomatic COVID-19 disease caused by variants of concerns (VoCs) in the BBIBP-CorV vaccine arm (s) compared to the control arm, 7 days after the second dose of study intervention.
Protection conferred by BBIBP-CorV vaccine against asymptomatic SARS-CoV-2 infection (any SARS-CoV-2 variant) | Till two years follow up from the date of enrollment
  Protection conferred by BBIBP-CorV vaccine against asymptomatic SARS-CoV-2 infection (any SARS-CoV-2 variant) measured as the reduction in incidence of RT-PCR-confirmed asymptomatic COVID-19 disease in the BBIBP-CorV vaccine arm (s) compared to the control arm 7 days after the second dose of study intervention.
Protection conferred by BBIBP-CorV vaccine against severe COVID-19 disease and COVID-19 associated death | Till two years follow up from the date of enrollment
  Protection conferred by BBIBP-CorV vaccine against severe COVID-19 disease and COVID-19 associated death, measured as the reduction in incidence of RT-PCR-confirmed severe COVID-19 hospitalization and death in the BBIBP-CorV vaccine arm (s) compared to the control arm.
Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in subset of participants | Till two years follow up from the date of enrollment
  Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in subset of participants, at Visit 2 (Day 0) , Visit 4 (day 28) , Visit 6 (day 56), Visit 7 (day 112), Visit 9 (day 140) Visit 10 (day 280) and Visit 11 (day 700)
Incidence of solicited adverse events, unsolicited adverse events and serious adverse events and adverse events of special interest (AESIs) in HIV-infected adults | Till two years follow up from the date of enrollment
  Incidence of local solicited adverse events within 7 days and systemic solicited adverse events within 14 days of each vaccination, unsolicited adverse events within 28 days of each vaccination, serious adverse events and adverse events of special interest (AESIs) according to Brighton Collaboration list for COVID-19 vaccine studies throughout the duration of the study in HIV-infected adults as compared to equal number of HIV-uninfected adults receiving the BBIBP-CorV vaccine and in HIV-infected adults receiving the control vaccine
Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in subset of participants in HIV-infected adults | Till two years follow up from the date of enrollment
  Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in subset of participants, at Visit 2 (Day 0) , Visit 4 (day 28) , Visit 6 (day 56), Visit 7 (day 112), Visit 9 (day 140) Visit 10 (day 280) and Visit 11 (day700) in HIV-infected adults as compared to in HIV-uninfected adults receiving the BBIBP-CorV vaccine and in HIV-infected adults receiving the control vaccine
SARS-CoV-2 sequence variants among HIV-infected and HIV-uninfected, BBIBP-CorV vaccine and placebo recipients | Till two years follow up from the date of enrollment
  SARS-CoV-2 sequence variants among HIV-infected and HIV-uninfected, BBIBP-CorV vaccine and placebo recipients
Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in the Arm 3 as compared to Arm 1 and 2 (subset participants). | Till two years follow up from the date of enrollment
  Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody in the Arm 3 as compared to Arm 1 and 2 (subset participants), at Visit 2 (Day 0) , Visit 4 (day 28) , Visit 6 (day 56), Visit 7 (day 112), Visit 9 (day 140) Visit 10 (day 280) and Visit 11 (day 700)
Incidence of adverse event (AE) after each vaccination, serious adverse event (SAE), adverse events of special interests (AESIs) according to Brighton Collaboration list for COVID-19 vaccine studies among participants receiving the study vaccines. | Till two years follow up from the date of enrollment
  Incidence of adverse event (AE) after each vaccination, serious adverse event (SAE), adverse events of special interests (AESIs) according to Brighton Collaboration list for COVID-19 vaccine studies throughout the duration of the study.
Humoral and cellular immune responses of HIV-infected participants as compared to HIV-uninfected vaccine and control arms (subset participants of Arms 1 and 2) | Till two years follow up from the date of enrollment
  Humoral and cellular immune responses of HIV-infected participants as compared to HIV-uninfected vaccine and control arms (subset participants of Arms 1 and 2) at Visit 2 (Day 0) , Visit 4 (day 28) , Visit 6 (day 56), Visit 7 (day 112), Visit 09 (day 140) Visit 10 (day 280) and Visit 11 (day 700).
Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody following booster dose of BBIBP-CorV vaccine | Till two years follow up from the date of enrollment
  Geometric Mean Titers (GMT) and Geometric Mean Fold Rise (GMFR) of anti-SARS-CoV-2 neutralizing antibody at Visit 7 (day 112), Visit 09 (day 140) Visit 10 (day 280) and Visit 11 (day 700) following booster dose of BBIBP-CorV vaccine.
Incidence of solicited adverse events, unsolicited adverse events and serious adverse events and adverse events of special interest (AESIs) among HIV uninfected adults. | Till two years follow up from the date of enrollment
  Incidence of local solicited adverse events within 7 days and systemic solicited adverse events within 14 days of booster dose, unsolicited adverse events within 28 days of booster dose and serious adverse events, and adverse events of special interest (AESIs) according to Brighton Collaboration list for COVID-19 vaccine studies throughout the duration of the study among HIV uninfected adults in the BBIBP-CorV vaccine arm (s) compared to the control arm.

OTHER OUTCOMES:
Acute phase reactants in COVID-19 patients that best predict COVID-19 disease and, hence, the control of protection against COVID-19 infection. | Till two years follow up from the date of enrollment
  Acute phase reactants in COVID-19 patients that best predict COVID-19 disease and, hence, the control of protection against COVID-19 infection.
Profile of the epitope-specific humoral immune response that tracks with protective immunity following natural infection or vaccine-induced immunity, using Systems Serology | Till two years follow up from the date of enrollment
  Profile of the epitope-specific humoral immune response that tracks with protective immunity following natural infection or vaccine-induced immunity, using Systems Serology
Any pregnancy outcomes after immunization in the intervention arm(s) as compared to control arm(s). | Till two years follow up from the date of enrollment
  Any pregnancy outcomes after immunization in the intervention arm(s) as compared to control arm(s)
The medical and psychological outcomes of COVID-19 patients in the first two years of follow-up | Till two years follow up from the date of enrollment
  The medical and psychological outcomes of COVID-19 patients in the first two years of follow-up
Identify novel SARS-CoV-2 host targets and host-virus interactions in low- and middle-income countries (LMIC) participants. | Till two years follow up from the date of enrollment
  Identify novel SARS-CoV-2 host targets and host-virus interactions in low- and middle-income countries (LMIC) participants.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marks, PhD, Principal Investigator — International Vaccine Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mozambique COVID-19 Situation — https://covid19.who.int/region/afro/country/mz